CLINICAL TRIAL: NCT06682026
Title: Mammography and Distraction Technique
Brief Title: Effect of Distraction Technique on Pain and Anxiety During Mammography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Dr., Hitit University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: mammography; Hitit Uni Non-Interventional (Registry Identifier: Ethics Committee)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Mammography Screening
Keywords: mammography; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): Written informed consent will be obtained from the patients immediately before they enter the procedure, and Personal Information Forms and the State Anxiety Inventory (STAI) will be administered to all participants. No intervention will be made to women in the control group. At the end of the procedure, the Visual Analog Scale (VAS) pain scale and the State Anxiety Inventory (STAI) will be applied to both groups.
- listening to music or chatting (Experimental): Written consent will be obtained from the patients just before they enter the procedure, and Personal Information Forms and the State Anxiety Inventory (STAI) will be applied to all participants.
  Women in the experimental group will be asked to listen to a lively music of their own choosing during the mammography, or for those who do not want music, their attention will be drawn in a different direction by chatting.
  At the end of the procedure, the Visual Acuity Scale (VAS) pain scale and the State Anxiety Inventory (STAI) will be applied to both groups.
  Interventions: Other: listening to music or chatting

INTERVENTIONS:
Other: listening to music or chatting — Written consent will be obtained from the patients just before they enter the procedure, and Personal Information Forms and the State Anxiety Inventory (STAI) will be applied to all participants.
  Women in the experimental group will be asked to listen to a lively music of their own choosing during the mammography, or for those who do not want music, their attention will be drawn in a different direction by chatting.
  At the end of the procedure, the Visual Acuity Scale (VAS) pain scale and the State Anxiety Inventory (STAI) will be applied to both groups.
  Arms: listening to music or chatting

SUMMARY:
One of the non-medical interventions aimed at reducing sensitization is the cognitive-behavioral approach, in which the individual's attention is shifted from a painful stimulus to an external stimulus. This non-pharmacological approach can be adopted to alleviate stress and reduce cortisol concentrations in response to stress. There are a limited number of studies in the literature using distraction techniques during mammography. This study will examine the effects of distraction techniques on pain and anxiety during mammography.

DETAILED DESCRIPTION:
According to global cancer statistics worldwide, breast cancer is the most commonly diagnosed cancer and the leading cause of cancer-related death in women. Breast cancer is the most common cancer among women in Turkey (40.7%). Early diagnosis of breast cancer reduces the mortality rate. Mammography is one of the important diagnostic tools used in breast cancer screening. Mammography is the most suitable method for screening with its easily accessible features and is the most successful imaging method in early diagnosis. The American Cancer Society recommends mammography for women aged 40-44. Women aged 45-54 should have mammography every year for breast cancer risk. The National Turkish Guide recommends that screening should start at age 40 and end at age 69 and be applied every two years (Özkan et al., 2016). However, studies show that most women do not routinely undergo mammography. The most important factor preventing mammography in women is defined as pain. Compression of the breasts during mammography is a necessary procedure to reduce radiation dose and improve image quality. Most women report experiencing pain during this compression procedure. Breast tenderness before mammography, family history of breast cancer, high level of education, carelessness of healthcare personnel performing mammography, and previous pain experience with mammography increase the level of pain during mammography. Although there are some techniques to relieve pain today, it is still important to find easier methods to apply. One of the non-medical interventions aimed at reducing sensitivity is the cognitive-behavioral approach; with this approach, the individual's attention is shifted from a painful stimulus to an external stimulus. This non-pharmacological approach can be adopted to alleviate stress and lower cortisol concentrations in response to stress.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-69,
* Those without a benign tumor in their breasts,
* Those without any hearing-related health problems.

Exclusion Criteria:

* Women under 40 and over 69,
* Women with suspected breast cancer.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 62 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 5 minutes after the procedure
  The Visual Analog Scale (VAS) is one of the most commonly used instruments to subjectively measure various states such as pain and anxiety. It is a 10 cm ruler with 0 at one end indicating no pain or anxiety and 10 at the other end indicating the worst imaginable pain or anxiety. The scale was used to assess pain after examination in only 2 groups.

SECONDARY OUTCOMES:
State Anxiety Inventory (STAI) | 5 minutes after the procedure
  To measure state anxiety, which refers to how one feels at the moment, and trait anxiety, which refers to how one feels in general. The State Anxiety Inventory consists of 20 self-reported 4-point Likert-type items, with negatively worded items reverse scored. Total scores range from 20 to 80, with higher scores indicating increased levels of anxiety.

IPD SHARING:
Plan to Share IPD: No